CLINICAL TRIAL: NCT02870972
Title: A Randomized, Double-blind, Placebo-controlled, Dose-ranging, Parallel-group Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BCX7353 as a Preventative Treatment to Reduce the Frequency of Attacks in Subjects With Hereditary Angioedema
Brief Title: Efficacy and Safety of BCX7353 to Prevent Angioedema Attacks in Subjects With Hereditary Angioedema
Acronym: APeX-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BCX7353-203
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part 1: BCX7353 350 mg once daily (Experimental): BCX7353 capsules, 350 mg dose administered once per day for 28 days
  Interventions: Drug: BCX7353
- Parts 2 and 3: BCX7353 250 mg once daily (Experimental): BCX7353 capsules, 250 mg dose administered once per day for 28 days
  Interventions: Drug: BCX7353
- Parts 2 and 3: BCX7353 125 mg once daily (Experimental): BCX7353 capsules, 125 mg dose administered once per day for 28 days
  Interventions: Drug: BCX7353
- Parts 1, 2 and 3: Placebo (Placebo Comparator): Placebo capsules, administered once per day for 28 days
  Interventions: Drug: Placebo
- Part 3: BCX7353 62.5 mg once daily (Experimental): BCX7353 capsules, 62.5 mg dose administered once per day for 28 days
  Interventions: Drug: BCX7353

INTERVENTIONS:
Drug: BCX7353 — Plasma kallikrein inhibitor
  Arms: Part 1: BCX7353 350 mg once daily; Part 3: BCX7353 62.5 mg once daily; Parts 2 and 3: BCX7353 125 mg once daily; Parts 2 and 3: BCX7353 250 mg once daily
Drug: Placebo
  Arms: Parts 1, 2 and 3: Placebo

SUMMARY:
This 3-part study will evaluate the safety and efficacy of an oral treatment, BCX7353, in preventing angioedema attacks in subjects with hereditary angioedema (HAE). In Part 1 of the study, eligible subjects will be randomized to receive oral BCX7353 or placebo for 4 weeks. Assuming successful completion of Part 1, additional subjects will be randomized in Part 2 to one of 2 lower doses of BCX7353 or placebo. Part 3 will enroll additional subjects into one of three doses of BCX7353 or placebo. The study will compare the number of acute attacks in each treatment group, as well as a number of other clinical and pharmacologic outcomes, and the safety and tolerability of each dose of BCX7353 compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* A clinical diagnosis of HAE type I or II
* Documented HAE attacks within a defined calendar period
* Access to acute attack medications
* Sexually active women of child-bearing potential and sexually active men must utilize effective contraception

Key Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Any clinical condition or medical history that would interfere with the subject's safety or ability to participate in the study
* Use of C1INH, androgens or tranexamic acid for prophylaxis of HAE attacks
* History of or current alcohol or drug abuse
* Infection with hepatitis B, hepatitis C or HIV
* Participation in any other investigational drug study currently or within the last 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emel Aygören-Pürsün, MD, Principal Investigator — University Hospital Frankfurt Goethe University
Locations (24):
- Australia (2):
  - Adelaide
  - Campbelltown
- Austria (2):
  - Graz
  - Vienna
- Canada (2):
  - Québec
  - Toronto
- Odense, Denmark
- Germany (3):
  - Berlin
  - Frankfurt
  - Ulm
- Budapest, Hungary
- Italy (3):
  - Milan
  - Padua
  - Salerno
- Skopje, North Macedonia
- Spain (3):
  - Barcelona
  - Madrid
  - Seville
- Zurich, Switzerland
- United Kingdom (5):
  - Brimingham
  - Bristol
  - London
  - Oxford
  - Southampton

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Farkas H, Balla Z. A review of berotralstat for the treatment of hereditary angioedema. Expert Rev Clin Immunol. 2023 Feb;19(2):145-153. doi: 10.1080/1744666X.2023.2150611. Epub 2022 Nov 29. PMID 36408587
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Aygoren-Pursun E, Bygum A, Grivcheva-Panovska V, Magerl M, Graff J, Steiner UC, Fain O, Huissoon A, Kinaciyan T, Farkas H, Lleonart R, Longhurst HJ, Rae W, Triggiani M, Aberer W, Cancian M, Zanichelli A, Smith WB, Baeza ML, Du-Thanh A, Gompels M, Gonzalez-Quevedo T, Greve J, Guilarte M, Katelaris C, Dobo S, Cornpropst M, Clemons D, Fang L, Collis P, Sheridan W, Maurer M, Cicardi M. Oral Plasma Kallikrein Inhibitor for Prophylaxis in Hereditary Angioedema. N Engl J Med. 2018 Jul 26;379(4):352-362. doi: 10.1056/NEJMoa1716995. PMID 30044938

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: HAE subjects attended a Screening Visit up to 21 days before the baseline visit, for assessment of eligibility to participate in the study.
Groups:
- Part 1: Berotralstat 350 mg: Berotralstat capsules, 350 mg dose administered once per day for 28 days
- Parts 2 & 3: Berotralstat 250 mg: Berotralstat capsules, 250 mg dose administered once per day for 28 days
- Parts 2 & 3: Berotralstat 125 mg: Berotralstat capsules, 125 mg dose administered once per day for 28 days
- Part 3: Berotralstat 62.5 mg: Berotralstat capsules, 62.5 mg dose administered once per day for 28 days
- Parts 1, 2 & 3: Placebo: Placebo capsules, administered once per day for 28 days
Period: Overall Study
Arm/Group | Part 1: Berotralstat 350 mg | Parts 2 & 3: Berotralstat 250 mg | Parts 2 & 3: Berotralstat 125 mg | Part 3: Berotralstat 62.5 mg | Parts 1, 2 & 3: Placebo
Started | 18 | 14 | 14 | 7 | 22
Completed | 17 | 14 | 14 | 7 | 22
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Berotralstat 350 mg | Parts 2 & 3: Berotralstat 250 mg | Parts 2 & 3: Berotralstat 125 mg | Part 3: Berotralstat 62.5 mg | Parts 1, 2 & 3: Placebo | Total
Number analyzed (Participants) | 18 | 14 | 14 | 7 | 22 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (11.6) | 40.9 (13.4) | 48.1 (12.6) | 38.9 (16.6) | 46.8 (11.1) | 44.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 10 | 6 | 13 | 46
  Male | 7 | 8 | 4 | 1 | 9 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 15 | 12 | 14 | 7 | 20 | 68
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Austria | 1 | 2 | 0 | 2 | 1 | 6
  Hungary | 1 | 0 | 0 | 0 | 2 | 3
  North Macedonia | 2 | 0 | 5 | 0 | 2 | 9
  Denmark | 1 | 0 | 3 | 1 | 3 | 8
  United Kingdom | 6 | 2 | 2 | 0 | 1 | 11
  Italy | 2 | 1 | 0 | 2 | 2 | 7
  Australia | 0 | 2 | 1 | 0 | 0 | 3
  Switzerland | 2 | 1 | 0 | 0 | 2 | 5
  Germany | 2 | 2 | 3 | 0 | 5 | 12
  Spain | 1 | 1 | 0 | 1 | 3 | 6
  France | 0 | 3 | 0 | 1 | 1 | 5
Adjusted qualifying HAE attack rate [Mean (Standard Deviation); unit: HAE attacks/week] | 0.84 (0.35) | 0.91 (0.43) | 0.94 (0.40) | 1.05 (0.44) | 0.87 (0.45) | 0.90 (0.41)

OUTCOME MEASURES:

1. Primary Outcome: Number of Confirmed HAE Attacks
Description: Efficacy was evaluated by the number of acute angioedema attacks. To ensure that consistent, objective assessments were used in accepting subject-reported attack data, a panel of expert physicians in the treatment of HAE patients adjudicated all subject-reported attacks prior to their inclusion in primary efficacy analyses.
Time Frame: Investigators collected data from patient diaries from the first day of dosing through to Day 29 or last day of dosing +24 hrs (the effective dosing period).
Population: The Full Analysis Set population included all subjects who were randomized, received at least 1 dose of study drug, and had post baseline HAE diary data recorded.
Measure: Least Squares Mean (Standard Error); unit: HAE attacks per week
Groups:
- Berotralstat 350 mg: Berotralstat capsules (350 mg) administered QD for 28 days
- Berotralstat 250 mg: Berotralstat capsules (250 mg) administered QD for 28 days
- Berotralstat 125 mg: Berotralstat capsules (125 mg) administered QD for 28 days
- Berotralstat 62.5 mg: Berotralstat capsules (62.5 mg) administered QD for 28 days
- Berotralstat: Berotralstat capsules administered QD for 28 days
- Placebo: Placebo capsules administered QD for 28 days
Arm/Group | Berotralstat 350 mg | Berotralstat 250 mg | Berotralstat 125 mg | Berotralstat 62.5 mg | Berotralstat | Placebo
Number analyzed (Participants) | 18 | 14 | 14 | 7 | 53 | 22
HAE attacks per week | 0.519 (0.115) | 0.527 (0.130) | 0.249 (0.130) | 0.852 (0.185) | 0.494 (0.067) | 0.952 (0.104)
Statistical Analysis 1: Comparison: Berotralstat vs Placebo; The primary analysis of treatment-effect was performed using an ANCOVA with the adjusted qualifying attack rate as the covariate; Test type: Superiority; p < 0.001, ANCOVA; Difference in Least Square Means = -0.458, 95% CI 2-sided [-0.703 to -0.214]
Statistical Analysis 2: Comparison: Berotralstat 350 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.006, ANCOVA; Difference in Least Square Means = -0.433, 95% CI 2-sided [-0.740 to -0.127]
Statistical Analysis 3: Comparison: Berotralstat 250 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.012, ANCOVA; Difference in Least Square Means = -0.425, 95% CI 2-sided [-0.755 to -0.095]
Statistical Analysis 4: Comparison: Berotralstat 125 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Difference in Least Square Means = -0.703, 95% CI 2-sided [-1.033 to 0.373]
Statistical Analysis 5: Comparison: Berotralstat 62.5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.639, ANCOVA; Difference in Least Square Means = -0.10, 95% CI 2-sided [-0.52 to 0.32]

2. Primary Outcome: Proportion of Subjects Who Were HAE Attack-free During the Entire Dosing Period
Description: Assessment of the proportion of subjects who had no HAE attacks during the entire dosing period
Time Frame: as for outcome 1
Population: The Full Analysis Set population included all subjects who were randomized, received at least 1 dose of study drug, and had post-baseline HAE diary data recorded.
Measure: Number; unit: participants
Arm/Group | Berotralstat 350 mg | Berotralstat 250 mg | Berotralstat 125 mg | Berotralstat 62.5 mg | Berotralstat | Placebo
Number analyzed (Participants) | 18 | 14 | 14 | 7 | 53 | 22
participants
  HAE Attack Free | 4 | 3 | 4 | 0 | 11 | 1
  HAE Attack Free (missing diary = attack) | 2 | 3 | 4 | 0 | 9 | 1
  HAE Attack Free (missing diary = exclude): number analyzed (Participants) | 14 | 13 | 14 | 7 | 48 | 22
  HAE Attack Free (missing diary = exclude) | 2 | 3 | 4 | 0 | 9 | 1
Statistical Analysis 1: Comparison: Berotralstat 350 mg vs Placebo; Test type: Superiority; p = 0.155, Fisher Exact; Difference vs placebo (%) = 17.7, 95% CI 2-sided [-3.4 to 38.8]
Statistical Analysis 2: Comparison: Berotralstat 250 mg vs Placebo; Test type: Superiority; p = 0.277, Fisher Exact; Difference vs placebo (%) = 16.9, 95% CI 2-sided [-6.3 to 40.1]
Statistical Analysis 3: Comparison: Berotralstat 125 mg vs Placebo; Test type: Superiority; p = 0.064, Fisher Exact; Difference vs placebo (%) = 24.0, 95% CI 2-sided [-1.2 to 49.2]
Statistical Analysis 4: Comparison: Berotralstat 62.5 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact; Difference vs placebo (%) = -4.5, 95% CI 2-sided [-13.2 to 4.2]
Statistical Analysis 5: Comparison: Berotralstat vs Placebo; Test type: Superiority; p = 0.097, Fisher Exact; Difference vs placebo (%) = -16.2, 95% CI 2-sided [-30.2 to -2.2]

3. Secondary Outcome: Number of Confirmed Abdominal HAE Attacks
Description: A prespecified secondary endpoint analyzed confirmed attacks by anatomical location; abdominal HAE attacks included any abdominal symptoms (i.e. swelling in the stomach/gut, or any symptoms of nausea, vomiting, or abdominal pain)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: HAE attacks per week
Arm/Group | Berotralstat 350 mg | Berotralstat 250 mg | Berotralstat 125 mg | Berotralstat 62.5 mg | Berotralstat | Placebo
Number analyzed (Participants) | 18 | 14 | 14 | 7 | 53 | 22
HAE attacks per week | 0.366 (0.073) | 0.324 (0.082) | 0.173 (0.083) | 0.404 (0.117) | 0.309 (0.042) | 0.370 (0.066)
Statistical Analysis 1: Comparison: Berotralstat vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.439, ANCOVA; Difference in Least Square Means = -0.061, 95% CI 2-sided [-0.216 to 0.094]
Statistical Analysis 2: Comparison: Berotralstat 350 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.968, ANCOVA; Difference in Least Square Means = -0.004, 95% CI 2-sided [-0.198 to 0.190]
Statistical Analysis 3: Comparison: Berotralstat 250 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.667, ANCOVA; Difference in Least Square Means = -0.045, 95% CI 2-sided [-0.254 to 0.164]
Statistical Analysis 4: Comparison: Berotralstat 125 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.065, ANCOVA; Difference in Least Square Means = -0.197, 95% CI 2-sided [-0.406 to 0.012]
Statistical Analysis 5: Comparison: Berotralstat 62.5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.797, ANCOVA; Difference in Least Square Means = 0.035, 95% CI 2-sided [-0.232 to 0.301]

4. Secondary Outcome: Number of Confirmed Peripheral HAE Attacks
Description: A prespecified secondary endpoint analyzed confirmed attacks by anatomical location; peripheral attacks included any with peripheral symptoms only (i.e. peripheral swelling or erythema marginatum).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: HAE attacks per week
Arm/Group | Berotralstat 350 mg | Berotralstat 250 mg | Berotralstat 125 mg | Berotralstat 62.5 mg | Berotralstat | Placebo
Number analyzed (Participants) | 18 | 14 | 14 | 7 | 53 | 22
HAE attacks per week | 0.160 (0.086) | 0.143 (0.097) | 0.098 (0.097) | 0.463 (0.138) | 0.179 (0.050) | 0.543 (0.078)
Statistical Analysis 1: Comparison: Berotralstat vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANOVA; Difference in Least Square Means = -0.364, 95% CI 2-sided [-0.547 to -0.181]
Statistical Analysis 2: Comparison: Berotralstat 350 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.001, ANCOVA; Difference in Least Square Means = -0.384, 95% CI 2-sided [-0.613 to -0.154]
Statistical Analysis 3: Comparison: Berotralstat 250 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.002, ANCOVA; Difference in Least Square Means = -0.401, 95% CI 2-sided [-0.647 to -0.154]
Statistical Analysis 4: Comparison: Berotralstat 125 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Difference in Least Square Means = -0.445, 95% CI 2-sided [-0.692 to -0.198]
Statistical Analysis 5: Comparison: Berotralstat 62.5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.614, ANCOVA; Difference in Least Square Means = -0.080, 95% CI 2-sided [-0.394 to 0.234]

5. Secondary Outcome: HAE Attacks Requiring Treatment
Description: A prespecified secondary endpoint analyzed the number of attacks requiring treatment with acute HAE medication (Berinert, Firazyr, Cinryze or Ruconest)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: HAE attacks per week
Arm/Group | Berotralstat 350 mg | Berotralstat 250 mg | Berotralstat 125 mg | Berotralstat 62.5 mg | Berotralstat | Placebo
Number analyzed (Participants) | 18 | 14 | 14 | 7 | 53 | 22
HAE attacks per week | 0.483 (0.109) | 0.449 (0.123) | 0.218 (0.1231) | 0.833 (0.174) | 0.450 (0.063) | 0.776 (0.098)
Statistical Analysis 1: Comparison: Berotralstat vs Placebo; The primary analysis of treatment-effect was performed using an ANCOVA with the terms of treatment and adjusted qualifying attack rate as the covariate; Test type: Superiority; p = 0.006, ANCOVA; Difference in Least Square Means = -0.326, 95% CI 2-sided [-0.557 to -0.095]
Statistical Analysis 2: Comparison: Berotralstat 350 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.047, ANCOVA; Difference in Least Square Means = -0.293, 95% CI 2-sided [-0.582 to 0.004]
Statistical Analysis 3: Comparison: Berotralstat 250 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.040, ANCOVA; Difference in Least Square Means = -0.327, 95% CI 2-sided [-0.638 to -0.016]
Statistical Analysis 4: Comparison: Berotralstat 125 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Difference in Least Square Means = -0.558, 95% CI 2-sided [-0.870 to -0.247]
Statistical Analysis 5: Comparison: Berotralstat 62.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.775, ANCOVA; Difference in Least Square Means = 0.057, 95% CI 2-sided [-0.339 to 0.454]

6. Secondary Outcome: HAE Disease Activity - Modified Angioedema Activity Score
Description: Activity of disease (i.e. disease severity) was assessed using a modified Angioedema Activity Score (AAS). The relevant endpoint for this study was the total modified AAS score, defined as the sum of the individual scores for 4 AAS domains (daily activities, appearance, physical discomfort, and overall severity) for all subject-reported attacks reported during the treatment period. Individual domain scores were based on answers to questions each of which had 4 possible responses scored 0-3 (0 - no impact; 1-3 - increasing levels of impact). The total modified AAS score per attack could range from 0 to 12; lower scores & higher scores represent lower & higher disease activities, respectively. However, the overall total modified AAS score reported for this study included the total scores for all subject-reported attacks, therefore the upper limit of the range was subject-specific. The statistical analysis of the total modified AAS scores for the treatment period is presented below.
Time Frame: 28-day treatment period + 1 day
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Berotralstat 350 mg | Berotralstat 250 mg | Berotralstat 125 mg | Berotralstat 62.5 mg | Placebo
Number analyzed (Participants) | 18 | 14 | 14 | 7 | 22
score on a scale | 14.070 (2.610) | 9.416 (2.952) | 7.256 (2.954) | 22.559 (4.200) | 18.519 (2.356)
Statistical Analysis 1: Comparison: Berotralstat 350 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.209, ANCOVA; Difference in Least Square Means = -4.449, 95% CI 2-sided [-11.453 to 2.555]
Statistical Analysis 2: Comparison: Berotralstat 250 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.019, ANCOVA; Difference in Least Square Means = -9.103, 95% CI 2-sided [-16.639 to -1.567]
Statistical Analysis 3: Comparison: Berotralstat 125 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.004, ANCOVA; Difference in Least Square Means = -11.263, 95% CI 2-sided [-18.808 to -3.718]
Statistical Analysis 4: Comparison: Berotralstat 62.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.405, ANCOVA; Difference in Least Square Means = 4.040, 95% CI 2-sided [-5.586 to 13.665]

7. Secondary Outcome: Angioedema Quality of Life (AE-QoL)
Description: Quality of Life (QoL) specific to hereditary angioedema (HAE) was assessed at baseline and Day 29 by a questionnaire (i.e. AE-QoL) consisting of 17 questions that spanned 4 domains (functioning, fatigue/mood, fear/shame, and nutrition). Each AE-QoL question had 5 answer options (scored 1-5), with lower and higher scores indicting less and more adverse impact, respectively. Per-subject scores for each domain were computed using the appropriate scoring algorithm applied to the question response scores for each domain. Per-subject total scores (including all 4 domains) were similarly computed using the question response scores for all 17 questions. The outputs from the scoring algorithm were normalized on a scale ranging from 0 (less adverse impact) to 100 (most adverse impact). The statistical analysis of the AE-QoL total score change from baseline to Day 29 is presented below.
Time Frame: The subject-completed AE-QoL was administered at baseline (Day 1) and at Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: AE-QoL score - change from baseline
Arm/Group | Berotralstat 350 mg | Berotralstat 250 mg | Berotralstat 125 mg | Berotralstat 62.5 mg | Placebo
Number analyzed (Participants) | 17 | 14 | 14 | 7 | 22
AE-QoL score - change from baseline | -12.59 (4.04) | -13.39 (4.44) | -28.95 (4.44) | -12.30 (6.32) | -4.47 (3.54)
Statistical Analysis 1: Comparison: Berotralstat 350 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.135, ANCOVA; Difference in Least Square Means = -8.12, 95% CI 2-sided [-18.826 to 2.584]
Statistical Analysis 2: Comparison: Berotralstat 250 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.121, ANCOVA; Difference in Least Square Means = -8.92, 95% CI 2-sided [-20.260 to 2.410]
Statistical Analysis 3: Comparison: Berotralstat 125 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, ANOVA; Difference in Least Square Means = -24.49, 95% CI 2-sided [-35.834 to -13.137]
Statistical Analysis 4: Comparison: Berotralstat 62.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.284, ANCOVA; Difference in Least Square Means = -7.84, 95% CI 2-sided [-22.316 to 6.640]

8. Secondary Outcome: DASS (Depression, Anxiety and Stress Scales)
Description: The Depression, Anxiety & Stress Scale (DASS) was used to measure the negative emotional states of depression, anxiety & stress. This assessment was based on a DASS questionnaire administered at baseline, Day 14 & Day 29. The questionnaire consisted of 3 DASS scales (depression, anxiety & stress) containing 14 items each on a scale of 0 to 3 (0, did not apply to me at all; 1, applied to me to some degree/some of the time; 2, applied to me to a considerable degree/a good part of the time; 3, applied to me very much or most of the time). Per-subject scores for the depression, anxiety & stress scales were obtained by summing the scores for the appropriate questionnaire items for the respective category. Total DASS scores were then derived as the sum of the 3 individual scales & ranged from 0 to 126. Higher & lower total scores are associated with more & less adverse impact, respectively. The statistical analysis of the total DASS score change from baseline to Day 29 is presented below.
Time Frame: The DASS was administered at baseline (Day 1), Day 14, and Day 29.
Population: The Full Analysis Set population included all subjects who were randomized, received at least 1 dose of study drug, and had post baseline HAE diary data recorded. Only data from subjects who completed the DASS-42 questionnaire (i.e. 3 DASS scales each containing 14 items) were included in this analyses. Data collected on the DASS-21 questionnaire were excluded.
Measure: Least Squares Mean (Standard Error); unit: DASS score - D29 change from baseline
Arm/Group | Berotralstat 350 mg | Berotralstat 250 mg | Berotralstat 125 mg | Berotralstat 62.5 mg | Placebo
Number analyzed (Participants) | 16 | 13 | 14 | 6 | 19
DASS score - D29 change from baseline | -7.627 (3.275) | -6.429 (3.609) | -10.840 (3.477) | -9.141 (5.336) | 0.643 (2.984)
Statistical Analysis 1: Comparison: Berotralstat 350 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.067, ANCOVA; Difference in Least Square Means = -8.270, 95% CI 2-sided [-17.132 to 0.592]
Statistical Analysis 2: Comparison: Berotralstat 250 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.136, ANCOVA; Difference in Least Square Means = -7.073, 95% CI 2-sided [-16.432 to 2.287]
Statistical Analysis 3: Comparison: Berotralstat 125 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.015, ANOVA; Difference in Least Square Means = -11.484, 95% CI 2-sided [-20.642 to -2.325]
Statistical Analysis 4: Comparison: Berotralstat 62.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.114, ANCOVA; Difference in Least Square Means = -9.785, 95% CI 2-sided [-22.001 to 2.431]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 1 of the study treatment period until 30 days after the last dose of study drug. Last dose was on study day 28 except in the event of early termination.
Arm/Group | Berotralstat 350 mg | Berotralstat 250 mg | Berotralstat 125 mg | Berotralstat 62.5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/14 | 0/14 | 0/7 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/14 | 0/14 | 0/7 | 0/22
Other Adverse Events (participants affected / at risk) | 14/18 | 11/14 | 7/14 | 4/7 | 15/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berotralstat 350 mg (N=18) | Berotralstat 250 mg (N=14) | Berotralstat 125 mg (N=14) | Berotralstat 62.5 mg (N=7) | Placebo (N=22)
Gastrointestinal infection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berotralstat 350 mg (N=18) | Berotralstat 250 mg (N=14) | Berotralstat 125 mg (N=14) | Berotralstat 62.5 mg (N=7) | Placebo (N=22)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 6 (6)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT02870972/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT02870972/SAP_001.pdf